CLINICAL TRIAL: NCT06029933
Title: Relative Vaccine Effectiveness of Adjuvanted Quadrivalent Inactivated Influenza Vaccine vs High-Dose Quadrivalent Inactivated Influenza Vaccine Among Adults ≥65 Years for the 2023-24 and 2024-25 Seasons
Brief Title: Fluad vs. Fluzone High-Dose Vaccine Effectiveness Among Adults ≥65 Years
Status: Recruiting | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Seqirus (Industry)
Responsible Party: Sponsor
Other Study IDs: 2033496
Record Dates: First submitted 2023-08-28; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Influenza; Community-acquired Pneumonia; Cardiovascular Events
MeSH Terms: conditions — Influenza, Human; Community-Acquired Pneumonia | interventions — fluad vaccine; Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fluad Recipients: Kaiser Permanente Northern California members aged ≥65 years who receive Adjuvanted Quadrivalent Inactivated Influenza Vaccine (aIIV4)
  Interventions: Biological: Adjuvanted Quadrivalent Inactivated Influenza Vaccine (aIIV4)
- Fluzone High-Dose Recipients: Kaiser Permanente Northern California members aged ≥65 years who receive High-Dose Quadrivalent Inactivated Influenza Vaccine (HD-IIV4)
  Interventions: Biological: High-Dose Quadrivalent Inactivated Influenza Vaccine (HD-IIV4)

INTERVENTIONS:
Biological: Adjuvanted Quadrivalent Inactivated Influenza Vaccine (aIIV4) — Fluad Quadrivalent vaccine is an inactivated influenza vaccine formulated to contain 60 mcg of hemagglutinin (HA) total, with 15 mcg from each of the four recommended influenza strains and the MF59 adjuvant in single-dose prefilled 0.5 mL syringes. Kaiser Permanente Northern California members ≥65 years may receive Fluad as part of routine clinical care during the influenza season.
  Other Names: Fluad
  Groups: Fluad Recipients
Biological: High-Dose Quadrivalent Inactivated Influenza Vaccine (HD-IIV4) — Fluzone High-Dose Quadrivalent vaccine is an inactivated split virion influenza vaccine formulated to contain 240 mcg of HA total, with 60 mcg from each of the four recommended influenza strains in single-dose prefilled 0.7 mL syringes. Kaiser Permanente Northern California members ≥65 years may receive Fluzone High-Dose as part of routine clinical care during the influenza season.
  Other Names: Fluzone High-Dose
  Groups: Fluzone High-Dose Recipients

SUMMARY:
This study will evaluate the relative vaccine effectiveness of quadrivalent adjuvanted inactivated influenza vaccine (aIIV4) versus quadrivalent high-dose inactivated influenza vaccine (HD-IIV4) in preventing polymerase chain reaction (PCR)-confirmed influenza and influenza-related outcomes in adults ≥65 years of age during the 2023/24 and 2024/25 influenza seasons. The study is an observational study conducted at Kaiser Permanente Northern California (KPNC), an integrated health care system in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years at the time of influenza vaccination
* KPNC member at the time of vaccination
* Receive either aIIV4 or HD-IIV4 at a KPNC facility during the 2023/24 and/or 2024/25 influenza seasons

Exclusion Criteria:

* Age <65 years at the time of influenza vaccination
* Received either aIIV4 or HD-IIV4 in the inpatient setting
* Receive more than one influenza vaccination during a single season period (i.e., 2023/24 or 2024/25 influenza seasons)
* Receive an influenza vaccination outside of KPNC

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study includes KPNC adults ≥65 years who receive Fluad or Fluzone High-Dose influenza vaccine as part of routine clinical care during the 2023/24 and/or 2024/25 influenza seasons.
Sampling Method: Non-Probability Sample
Enrollment: 960000 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
PCR-confirmed influenza | ≥14 days after vaccination until date of outcome, death, loss-to-follow-up, or end of each season (estimated May 2024 or May 2025)
  KPNC members ≥65 years who receive Fluad or Fluzone High-Dose will be retrospectively assessed for the presence of PCR-confirmed influenza. This outcome will be assessed in single-season analyses (2023/24 and 2024/25 separately) and a pooled 2-seasons analysis (2023/24 and 2024/25 combined).

SECONDARY OUTCOMES:
Emergency department visit or hospitalization for PCR-confirmed influenza | ≥14 days after vaccination until date of outcome, death, loss-to-follow-up, or end of each season (estimated May 2024 or May 2025)
  KPNC members ≥65 years who receive Fluad or Fluzone High-Dose will be retrospectively assessed for an emergency department visit or hospitalization for PCR-confirmed influenza. This outcome will be assessed in single-season analyses (2023/24 and 2024/25 separately) and a pooled 2-seasons analysis (2023/24 and 2024/25 combined).
Hospitalization for PCR-confirmed influenza | ≥14 days after vaccination until date of outcome, death, loss-to-follow-up, or end of each season (estimated May 2024 or May 2025)
  KPNC members ≥65 years who receive Fluad or Fluzone High-Dose will be retrospectively assessed for hospitalization for PCR-confirmed influenza. This outcome will be assessed in a pooled 2-seasons analysis (2023/24 and 2024/25 combined).
Hospitalization for all-cause community-acquired pneumonia | ≥14 days after vaccination until date of outcome, death, loss-to-follow-up, or end of each season (estimated May 2024 or May 2025)
  KPNC members ≥65 years who receive Fluad or Fluzone High-Dose will be retrospectively assessed for hospitalization for all-cause community-acquired pneumonia. This outcome will be assessed in single-season analyses (2023/24 and 2024/25 separately) and a pooled 2-seasons analysis (2023/24 and 2024/25 combined).

OTHER OUTCOMES:
Hospitalization for cardiovascular events | ≥14 days after vaccination until date of outcome, death, loss-to-follow-up, or end of each season (estimated May 2024 or May 2025)
  KPNC members ≥65 years who receive Fluad or Fluzone High-Dose will be retrospectively assessed for hospitalization for cardiovascular events. This outcome will be assessed in single-season analyses (2023/24 and 2024/25 separately) and a pooled 2-seasons analysis (2023/24 and 2024/25 combined).
PCR-confirmed influenza in subgroups with comorbidities | ≥14 days after vaccination until date of outcome, death, loss-to-follow-up, or end of each season (estimated May 2024 or May 2025)
  KPNC members ≥65 years with comorbidities (e.g., cardiovascular and respiratory conditions, diabetes, obesity) who receive Fluad or Fluzone High-Dose will be retrospectively assessed for hospitalization for PCR-confirmed influenza. This outcome will be assessed in a pooled 2-seasons analysis (2023/24 and 2024/25 combined).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Northern California (entire region), Oakland, California, United States